CLINICAL TRIAL: NCT04838327
Title: Rare Subtypes of Gastrointestinal Cancers - Real-world Data and Liquid Biopsies
Brief Title: Rare Subtypes of Gastrointestinal Cancers
Status: Recruiting | Type: Observational
Sponsor: Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Louise Bach Callesen, MD, Aarhus University Hospital
Other Study IDs: 1-10-72-7-21
Record Dates: First submitted 2021-04-01; First posted 2021-04-09 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Cancer of Gastrointestinal Tract
MeSH Terms: conditions — Gastrointestinal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A single-arm prospective observational translational study of biomarkers in patients receiving targeted treatment for rare subtypes of cancer of the Gastrointestinal Tract.

DETAILED DESCRIPTION:
In this study, the investigators seek to investigate biological aspects in patients receiving targeted treatment for rare subtypes of cancer of the Gastrointestinal.

The targeted treatment will be given as per standard of care. Translational blood samples will be drawn pre-treatment, before the third cycle of chemotherapy, and hereafter corresponding to the planned imaging during treatment and follow up.

The total cell free DNA will be quantified in all samples. The samples will be analyzed for tumor specific mutations such as the KRAS, BRAF, and NRAS oncogenes, by ddPCR. Circulating tumor DNA will also be identified by hypermethylation markers, and a focused panel of next generation sequencing can be applied. The samples will also be analyzed for immune-related biomarkers.

The investigators expect to include up to 130 patients.

This is a purely observational translational study. Results will be analysed in relation to outcome data.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of a rare subtype of GI cancer including BRAF V600E mutation, MSI-H, HER2 and others
* Diagnosis of cancer of the gastrointestinal tract may be made by histo- or cyto-pathology, or by clinical and imaging criteria
* Planned for targeted treatment
* Age 18 years or older
* Able to understand written information
* Consent to samples for translational research

Exclusion Criteria:

* Conditions precluding translational blood sampling
* Another concomitant cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of patients with rare subtypes of cancer of the gastrointestinal tract, who by standard of care are candidates for targeted treatment
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2021-08-16 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility and translational analysis | 2 years last patient
  Investigating potential prognostic and predictive markers for efficacy by molecular characteristics and mutational analysis. We seek to describe the prognostic and predictive value of cfDNA, ctDNA and other markers, e.g. evaluate baseline cf- and ctDNA levels, fluctuations of cf- and ctDNA during treatment and follow up.

SECONDARY OUTCOMES:
Response rate | 6 months post-treatment
  According to RECIST version 1.1
Progression Free Survival | 2 years last patient
  Time from inclusion to progression according to RECIST version 1.1
Overall Survival | 2 years last patient
  Time from inclusion til death from any cause
Quality of Life by EORTC QLQ-C30 | 2 years last patient
  Patients are asked to indicate their symptoms during the past week(s). Scores can be linearly transformed to provide a score from 0 to 100. Higher scores represent better functioning on the functional scales and a higher level of symptoms on the symptom scales.

CONTACTS AND LOCATIONS:
Overall Officials: Louise B Callesen, MD, Principal Investigator — Experimental Clinical Oncology
Locations (1):
- Department of Oncology, Aarhus University Hospital, Aarhus N, Denmark

IPD SHARING:
Plan to Share IPD: No